CLINICAL TRIAL: NCT03387332
Title: A Phase I Study of the Safety, Pharmacokinetic and Pharmacodynamic Properties of Intravenously Administered APG-1252 in Patients With Small Cell Lung Cancer (SCLC) or Advanced Solid Tumors.
Brief Title: APG-1252 in Patients With SCLC or Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The company adjusts strategy.
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-1252-CH-001
Record Dates: First submitted 2017-12-13; First posted 2018-01-02 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Small Cell Lung Cancer and Other Solid Tumors
Keywords: Bcl-2/Bcl-xL dual inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pelcitoclax; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APG-1252 (Experimental): The starting dose for this study was 40 mg and 1 patient would be enrolled at this dose level. The dose escalation will convert to a standard 3+3 design following the occurrence of DLT or two ≥ Grade 2 adverse event or at doses 80 mg.
  Interventions: Drug: APG-1252

INTERVENTIONS:
Drug: APG-1252 — Multiple dose cohorts, 30 minute IV infusion, twice weekly for 3 weeks of a cycle with 28 days.
  Other Names: APG-1252 for injection

SUMMARY:
APG-1252 is a highly potent Bcl-2 family protein inhibitor, a promising drug candidate which shown high binding affinities to Bcl-2, Bcl-xL and Bcl-w. The preclinical studies have shown that APG-1252 alone achieves complete and persistent tumor regression in multiple tumor xenograft models with a twice weekly or weekly dose-schedule, including SCLC, colon, breast and ALL cancer xenografts; achieves strong synergy with the chemotherapeutic agents, indicating that APG-1252 may have a broad therapeutic potential for the treatment of human cancer as a single agent and in combination with other classes of anticancer drugs. APG-1252 is intended for the treatment of patients with SCLC or other solid tumors. Upon completion of the Phase 1 dose escalation study to establish the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and/or recommended phase 2 dose (RP2D), several phase Ib/II studies will be implemented accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed small cell lung cancer (SCLC) or other solid tumors;
2. Male or non-pregnant, non-lactating female patients age ≥18 years;
3. Locally advanced or metastatic disease for which no standard therapy is judged appropriate by the investigator;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2;
5. Adequate hematologic function as indicated by:

   1. Platelet count ≥ 100,000/mm3
   2. Hemoglobin ≥ 9.0g/dL
   3. Absolute neutrophil count (ANC) ≥1000/µL
6. Adequate renal and liver function as indicated by:

   1. Serum creatinine ≤ 1.5 x upper limit of normal (ULN); if serum creatinine is >1.5 X ULN, creatinine clearance must be ≥ 50 mL/min (see Section 22.3).
   2. Total bilirubin ≤1.5 x ULN; If Gilbert's Syndrome may have Bilirubin> 1.5 x ULN
   3. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤3 x ULN of institution's normal range; for patients with known liver metastases, AST and ALT may be ≤ 5 x ULN.
   4. Coagulation: aPTT and PT<1.2 x the upper limit of normal
7. Brain metastases with clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function & no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.
8. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug;
9. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures);
10. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Receiving concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, with the exception of hormones for hypothyroidism or estrogen replacement therapy (ERT), anti estrogen analogs, agonists required to suppress serum testosterone levels); or any investigational therapy, or has had tumor embolization or tumor lysis syndrome (TLS) within 14 days prior to the first dose of study drug.
2. Steroid therapy for anti-neoplastic intent within 7 days prior to the first dose of study drug.
3. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to < Grade 2;
4. Known bleeding diathesis/disorder;
5. Recent history of non-chemotherapy induced thrombocytopenia associated bleeding within 1 year prior to first dose of study drug.
6. Have active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
7. Serious gastrointestinal bleeding within 3 months;
8. Use of therapeutic doses of anti-coagulants is excluded, along with anti-platelet agents; low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter are permitted.
9. Received a biologic (G-CSF, GM-CSF or erythropoietin) within 28 days prior to the first dose of study drug.
10. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry;
11. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry.
12. Neurologic instability per clinical evaluation due to tumor involvement of the central nervous system (CNS). Patients with CNS tumors that have been treated, are asymptomatic and who have discontinued steroids (for the treatment of CNS tumors) for >28 days may be enrolled;
13. Active symptomatic fungal, bacterial and/or viral infection including, but not limited to, active human immunodeficiency virus (HIV) or viral hepatitis (B or C);
14. Diagnosis of fever and neutropenia within 1 week prior to study drug administration.
15. Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
16. Prior treatment with Bcl-2/Bcl-xL inhibitors.
17. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Dose limit toxicity (DLT) determination | 18-24 months
  Number of participants with APG-1252 treatment-related adverse events as assessed by CTCAE v4.03
Maximum tolerated dose (MTD) determination | 18-24 months
  If ≥ 2/6 patients develop a DLT at any dose level, then this dose will be declared as the MTD.

SECONDARY OUTCOMES:
Pharmacokinetic evaluation | 18-24 months
  Peak plasma concentration (Cmax) will be assessed on all participants with APG-1252 treatments.
Preliminary efficacy assessment | 18-24 months
  Patients will be evaluated for response every 2 cycles (i.e., 8 weeks), according to the new response evaluation criteria in solid tumors: revised RECIST Guideline, Version 1.1

OTHER OUTCOMES:
Pharmacokinetic evaluation | 18-24 months
  Area under the plasma concentration versus time curve (AUC) will be assessed on all participants with APG-1252 treatments
Pharmacodynamic evaluation | 18-24 months
  Apoptosis will be assessed on the patients treated with APG-1252

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, M.D., Ph.D., Study Director — Ascentage (Suzhou) Pharma Group Inc
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China